CLINICAL TRIAL: NCT02784574
Title: Follow-up After Intensive Care Treatment: a Questionnaire Survey of Intensive Care Aftercare in Denmark.
Brief Title: Post ICU Follow up: A Questionnaire Survey of Aftercare in Denmark
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CK1-Survey
Record Dates: First submitted 2016-04-20; First posted 2016-05-27 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Critical Illness; Intensive Care Unit Syndrome
Keywords: Rehabilitation; Aftercare
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to investigate current aftercare activities in Denmark after intensive care unit (ICU) treatment. The hypothesis is that a large number of hospitals offer aftercare, and these interventions are heterogenic and differ between hospitals and regions.

This study is an electronic questionnaire survey that aim to describe and map Danish aftercare activities, and future development plans in this field.

DETAILED DESCRIPTION:
Annually, more than 30,000 patients are admitted for treatment at Danish intensive care units (ICUs). These critically ill patients are some of the most vulnerable in the health care system.

For years, focus has primarily been on treatment and survival of this patient group. As treatment effectiveness has gradually increased, the overall survival rate is now above 80%. Consequently, the period following ICU discharge has gained increasing focus and follow up interventions in the period after ICU treatment have become more common. These different follow up interventions has given name to the concept of 'aftercare'. Aftercare activities includes both early rehabilitation initiated during the continued hospital admission and also the following rehabilitation after hospital discharge.

Complications after intensive care treatment are numerous, including both physical, cognitive and psychological impairments, e.g. depression, muscle weakness, anxiety and social isolation. Together these symptoms are defined as post intensive care syndrome (PICS).

While it is clear that a need for aftercare exists, the optimal evidence based activities remains to be determined. The current follow-up activities are established as local initiatives and the methods vary greatly. Examples of present aftercare interventions include use of diaries, follow-up consultations, revisiting the ICU and assessment of quality of life.

A recent systematic review examined these different rehabilitation efforts, without finding significant effects of the present interventions, although usage of ICU-diaries had a minor preventive effect on post-traumatic stress syndrome (PTSD). A Danish meta-analysis from 2015 on follow-up consultations showed similar results.

Aftercare is a rapidly developing area and it is necessary to further investigate this important topic. Therefore, the investigators want to describe the current level of aftercare with a new mapping of activities in all Danish ICUs. Hereby, the investigators hope to create a better and up-to-date foundation for further development within Danish aftercare. Furthermore, the investigators wish to research on the clinician-experienced (the participants) attitude towards and limitations for aftercare activities, in order to discuss directions for future development.

ELIGIBILITY:
Inclusion Criteria:

* All Intensive Care Units in Denmark treating adult patients.

Exclusion Criteria:

Intensive care units with a specialty field within these four groups:

* Neurology and neurosurgery
* Cardiothoracic surgery
* Pediatrics or neonatology (PICU/NICU)
* Postoperative care units

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Intensive Care Units in Denmark treating adult patients.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of ICUs offering early aftercare to patients after discharge from ICU | From May 15th to September 31st 2016
  The respondent will choose 'yes' or 'no'
Incidence of ICUs offering late aftercare to patients after discharge from hospital | From May 15th to September 31st 2016
  The respondent will choose 'yes' or 'no'

SECONDARY OUTCOMES:
Size of hospital (number of beds) | From May 15th to September 31st 2016
Size of ICU (number of beds) | From May 15th to September 31st 2016
Early aftercare: Use of protocol or checklist at patient visit | From May 15th to September 31st 2016
  The respondent will choose 'yes' or 'no'
Late aftercare: Use of protocol or checklist at patient visit | From May 15th to September 31st 2016
  The respondent will choose 'yes' or 'no'
Early aftercare: Selection of patients offered aftercare | From May 15th to September 31st 2016
  The respondent will choose from a list of options: All patients, Depending of length of stay, days with mechanical ventilation, or other: the respondent will specify
Late aftercare: Selection of patients offered aftercare | From May 15th to September 31st 2016
  The respondent will choose from a list of options: All patients, Depending of length of stay, days with mechanical ventilation, or other: the respondent will specify
Early aftercare: Time from ICU-discharge to first contact | From May 15th to September 31st 2016
  The respondent will choose from a list of options: How many hours to days until the patient is contacted at the general wards
Late aftercare: Time from hospital discharge to first contact | From May 15th to September 31st 2016
  The respondent will choose from a list of options: How many months from discharge, until the patient is contacted
Early aftercare: Aftercare team members | From May 15th to September 31st 2016
  The respondent will choose from a list of options: The personnel participating in the aftercare: Doctor, nurse, occupational therapist, physical therapist, pharmacist, psychologist or other
Early aftercare: Consumption of time | From May 15th to September 31st 2016
  The respondent will choose from a list of options: How much time is spent (in minutes) pr. contact with the patient
Late aftercare: Aftercare team members | From May 15th to September 31st 2016
  The respondent will choose from a list of options: The personnel participating in the aftercare: Doctor, nurse, occupational therapist, physical therapist, pharmacist, psychologist or other
Late aftercare: Consumption of time | From May 15th to September 31st 2016
  The respondent will choose from a list of options: How much time is spent (in minutes) pr. contact with the patient
Early aftercare: Type of aftercare interventions during general ward stay | From May 15th to September 31st 2016
  The respondent will be choosing interventions from a list, and also be able to specify other interventions not present on the list
Late aftercare: Type of aftercare interventions after hospital discharge | From May 15th to September 31st 2016
  The respondent will be choosing interventions from a list, and also be able to specify other interventions not present on the list
Early aftercare: Type of screening tools or other methods used for patient assessment | From May 15th to September 31st 2016
  The respondent will be choosing screening tools and methods from a list, and also be able to specify other screening tools and methods not present on the list
Late aftercare: Type of screening tools or other methods used for patient assessment | From May 15th to September 31st 2016
  The respondent will be choosing screening tools and methods from a list, and also be able to specify other screening tools and methods not present on the list
Late aftercare: Contact method | From May 15th to September 31st 2016
  The respondent will choose from a list of options: How the ICU contacts the patient after hospital discharge. By phone, by letter, by mail, by digital inbox
Late aftercare: Participation of family members | From May 15th to September 31st 2016
  The respondent will choose from a list: Whether the family is invited to participate in the consultation with the patient or not. Yes/No
Classifications of reasons for not having an aftercare programme at ICUs without an aftercare programme | From May 15th to September 31st 2016
  The respondent will choose from a list of options: Not enough money, resistance from the general wards, not an important subject, and also be able to write their own answer.
The responsible party for the financing of aftercare | From May 15th to September 31st 2016
  The respondent will choose from a list of options: The ICU itself, the general ward, the region or through funds?
The respondent's own assessment of how aftercare will be prioritized at their ICU in one year. | From May 15th to September 31st 2016
  The respondent will choose on a scale: More aftercare? Same level of aftercare? Less aftercare?
Should aftercare be offered? | From May 15th to September 31st 2016
  The respondent will choose on a scale: Totally agree, partially agree, neither agree or disagree, partially disagree, totally disagree

CONTACTS AND LOCATIONS:
Overall Officials: Cilia KW Kjer, Bach.med, Principal Investigator — Køge Hospital
Locations (1):
- Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haggstrom M, Asplund K, Kristiansen L. How can nurses facilitate patient's transitions from intensive care?: a grounded theory of nursing. Intensive Crit Care Nurs. 2012 Aug;28(4):224-33. doi: 10.1016/j.iccn.2012.01.002. Epub 2012 Mar 3. PMID 22386583
- [Background] Broomhead LR, Brett SJ. Clinical review: Intensive care follow-up--what has it told us? Crit Care. 2002 Oct;6(5):411-7. doi: 10.1186/cc1532. Epub 2002 Aug 15. PMID 12398780
- [Background] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Wolters A, Bouw M, Vogelaar J, Tjan D, van Zanten A, van der Steen M. The postintensive care syndrome of survivors of critical illness and their families. J Clin Nurs. 2015 Mar;24(5-6):876-9. doi: 10.1111/jocn.12678. Epub 2014 Dec 1. No abstract available. PMID 25441007
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Mehlhorn J, Freytag A, Schmidt K, Brunkhorst FM, Graf J, Troitzsch U, Schlattmann P, Wensing M, Gensichen J. Rehabilitation interventions for postintensive care syndrome: a systematic review. Crit Care Med. 2014 May;42(5):1263-71. doi: 10.1097/CCM.0000000000000148. PMID 24413580
- [Background] Jensen JF, Thomsen T, Overgaard D, Bestle MH, Christensen D, Egerod I. Impact of follow-up consultations for ICU survivors on post-ICU syndrome: a systematic review and meta-analysis. Intensive Care Med. 2015 May;41(5):763-75. doi: 10.1007/s00134-015-3689-1. Epub 2015 Mar 3. PMID 25731633
- [Background] Egerod I, Risom SS, Thomsen T, Storli SL, Eskerud RS, Holme AN, Samuelson KA. ICU-recovery in Scandinavia: a comparative study of intensive care follow-up in Denmark, Norway and Sweden. Intensive Crit Care Nurs. 2013 Apr;29(2):103-11. doi: 10.1016/j.iccn.2012.10.005. Epub 2013 Jan 20. PMID 23340012
- [Background] Engstrom A, Andersson S, Soderberg S. Re-visiting the ICU Experiences of follow-up visits to an ICU after discharge: a qualitative study. Intensive Crit Care Nurs. 2008 Aug;24(4):233-41. doi: 10.1016/j.iccn.2008.03.002. Epub 2008 Apr 22. PMID 18434156
- [Background] Van Der Schaaf M, Bakhshi-Raiez F, Van Der Steen M, Dongelmans DA, De Keizer NF. Recommendations for intensive care follow-up clinics; report from a survey and conference of Dutch intensive cares. Minerva Anestesiol. 2015 Feb;81(2):135-44. Epub 2014 May 14. PMID 24824957
- See also: Database DI. DID's - Alle mortalitetsmål. 2014 1-10. — https://www.sundhed.dk/sundhedsfaglig/kvalitet/kliniske-kvalitetsdatabaser/specifikke-procedurer/intensiv-database/